CLINICAL TRIAL: NCT04027660
Title: Volumetric (Hard and Soft Tissue) Alterations in Immediate Zirconia Implants
Brief Title: Outcome of Immediate Zirconia Implants
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Implantology Institute (Other)
Responsible Party: Principal Investigator, Andre Chen, Assistant Professor, Implantology Institute
Other Study IDs: II-10
Record Dates: First submitted 2019-07-12; First posted 2019-07-22 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Implant
Keywords: dentistry; zirconia; implants

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed Immediate Zirconia Implants: Group Formation : patients that require a tooth extraction and have the following clinical indications to be enrolled in an immediate implant.
  1. No Active Infection
  2. No loss of buccal plate
  3. ASA 1 or ASA 2 Patient
  Extraction of the tooth will be performed and in the same clinical act, a zirconia dental implant will be placed toghether with a provisional or an individualized customs healing abutment. The jumping gap will be filled with a xenograft biomaterial.
  Final Zirconia Crown delivered 3 month after healing.
  3 STL files will be generated - Before extraction, at Final impression level 3 month after implant placement, at 3 month after final prosthesis insertion
  Measure 1,2 and 3 will be at the gingival margin(measure 1), at 2mm (measure 2) and 4 mm (measure 3) apical to gingival margin. Both palatal and buccal references are joined by a line that gives a distance.Difference on the dimensions of each line with different time of evaluation represent ridge loss.
  Interventions: Device: Immediate Zirconia Dental Implant
- Non-exposed delayed Zirconia implants: Group Formation : patients that require a tooth extraction and have the following clinical indications not to be enrolled in an immediate implant.
  1. Active Infection
  2. Loss of the buccal plate.
  Extraction will be performed but a classical implant approach will be made, that include a waiting period of 3 month before implant placement and 3 month after osseointegration period before place final crown.
  Implant placement with Guided bone regeneration (xenograft), if needed. Final Zirconia Crown 3 month after implant placement.
  4 STL files will be generated - Before extraction, before implant placement, at Final impression level 3 month after implant placement, at 3 month after final prosthesis insertion
  Measure 1,2 and 3 the same has the other group

INTERVENTIONS:
Device: Immediate Zirconia Dental Implant — For the Exposed Group the Intervention will be the following
  The Surgical procedure will envolve :
  1. Administration of Articain 1:200.000
  2. No flap procedure
  3. Place a Zirconia Implant on the alveolar post extraction socket
  4. Place xenograft biomaterial in the jumping gap
  5. Place a provisional crown/individualized healing abutment
  The Prosthodontic procedure will evolve:
  * Final Impression with a IOS
  * Placement of the Final Crown
  * 3 month post crown post op
    3 IOS will be made for volumetric evaluation :
    1. before tooth extraction
    2. 3 month of Osseointegration for final impression
    3. 3 month after final crown is placed
  Final STL evaluation will be performed on a specialized software for volumetric measurements
  Groups: Exposed Immediate Zirconia Implants

SUMMARY:
The aim is to study bone and soft tissue response to zirconia immediate implants.Volumetric changes will be measured before tooth extraction and after final crow placement.

DETAILED DESCRIPTION:
Bone remodeling around immediate implants is a reality in clinical and literature arena. much is known about titanium implants but little in zirconia implants

In patients that require a tooth extraction anywhere in the oral cavity except 3rd molars are candidates fo the study. Once clinical conditions are establish and medical clearance is ok, the decision for an immediate implant is taken.

Patient will undergo for an intraoral Scanner (IOS, Trios 3Shape) to get an STL file of the previous situation.

On the day of surgery an atraumatically tooth extraction is performed (without rasing a flap) and a Zirconia implant is inserted on the alveolar socket.

The jumping gap (distance from crystal bone to implant body will be filled with a zenograft type of biomaterial) no sutures or membrane will be used.

A provisional crown or an individualized healing abutment will be placed. After 3 month healing an IOS will be made for crown fabrication and a second STL file generated.

After 15 days final crown will be placed, and 3 month after a 3rd IOS made to get the 3rd and final STL file.

An STL software will then make the correlation between the volume behavior in those 3 stages.

The control group, patients go for tooth extraction but no immediate implant and undergo with a classic protocol for implant placement. In this case the STL files are taken pre-operatory, before implant placement 3 month after tooth extraction, 2 month after implant placement (at final impression level), and 3 month after crown placement.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a non-restorable tooth schedule for extraction
2. Anywhere on the mouth except 3rd molar teeth
3. Tooth site with no active infection
4. No loss of the buccal, palatal or inter proximal bone
5. If chronical apical pathology, the six should be less that 4 mm diameter
6. ASA 1 or ASA 2 Patient
7. Sings the Informed consent -

Exclusion Criteria:

1. Site has an active infection
2. Periapical lesion Beyond 5 mm
3. Bone resorption of buccal, palatal or inter proximal plate beyond 2 mm
4. Patient doesn't want an immediate implant
5. Patient doesn't want a Zirconia Implant
6. ASA 3 or ASA 4 Patient
7. Refuse to Sign informed consent -

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sequential recruiting, middle age, moderate to high income
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2019-01-26 (Actual); Primary Completion 2020-07-26 (Estimated); Study Completion 2020-08-26 (Estimated)

PRIMARY OUTCOMES:
Ridge dimensions (Bone and soft tissue from buccal to palatal) Changes from Implant placement in alveolar extraction sockets (Day 1) to final impression, 2 month after osseointegration (Day 2), in Zirconia Immediate Implants | 1 year
  Physiologic resorption rate (measured in a buccal to palatal dimension) from day 1 - Immediate implant in an alveolar extraction socket to Day 2 - Day of final Impression measured by STL superimposition. Acquisition of STL File with an IOS in both time frames, and in a STL reader software (Geomagic Control X) we merge them with the corresponding common landmarks for a best fit alignment.
  Measure include, Total bone and soft tissue volume loss (in cubic centimeters). Bone collapse measured in mm from the most buccal point to most palatal point of the ridge.
Ridge dimensions (Bone and soft tissue from buccal to palatal) Changes from final impression (Day 2 ) to 2 month after osseointegration (Day 3), in Zirconia Immediate Implants | 1Year
  Physiologic resorption rate from Day 2 - Day of final Impression to Day 3- 3 month after final crown insertion measured by STL superimposition. Acquisition of STL File with an IOS in both time frames, and in an STL reader software (Geomagic Control X) we merge them with the corresponding common landmarks for a best fit alignment.
  Measure include, Total bone and soft tissue volume loss (in cubic centimeters). Bone collapse measured in mm from the most buccal point to most palatal point of the ridge.
Ridge dimensions (Bone and soft tissue from buccal to palatal) Changes from Implant placement in alveolar extraction sockets (Day 1) to 2 month after osseointegration (Day 3), in Zirconia Immediate Implants | 1year
  Physiologic resorption rate from Day 1 - implant placement to Day 3- 3 month after final crown insertion measured by STL superimposition. Acquisition of STL File with an IOS in both time frames, and in an STL reader software (Geomagic Control X) we merge them with the corresponding common landmarks for a best fit alignment.
  Measure include, Total bone and soft tissue volume loss (in cubic centimeters). Bone collapse measured in mm from the most buccal point to most palatal point of the ridge.

SECONDARY OUTCOMES:
Survival Rate of Zirconia Immediate implants | 5 years
  Evaluate osseoitegration and the long term behavior of immediacy with zirconia implants
Rate of complications | 1 Year
  Track a log book on complications when using immediate zirconia implants

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Implantologia, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No